CLINICAL TRIAL: NCT01427166
Title: Evaluation of Non Invasive Imaging for Assessing the Pathophysiology of Cording in Patients Treated for Breast Cancer
Brief Title: Non-Invasive Imaging for Cording in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alphonse Taghian, MD, PhD, Chief of Breast Service, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-279; R01CA139118 (NIH)
Record Dates: First submitted 2011-08-25; First posted 2011-09-01 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Cording; Lymphedema; upper extremity cording; following treatment
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ultrasound imaging (Experimental): Cords that are present in the participant's axilla and/or arm will be imaged with an ultrasound
  Interventions: Other: Non invasive venous ultrasound

INTERVENTIONS:
Other: Non invasive venous ultrasound — Subjects will undergo a venous duplex ultrasound, on a General Electric LOGIQ-9 unit with a Phillips-IU-22 probe

SUMMARY:
To date, the scientific literature has yet to provide sufficient evidence regarding the pathophysiology of cording. The objective of this protocol is to evaluate the utility of non invasive vascular imaging for assessing the pathophysiology of cording in a small study cohort of patients who were treated for breast cancer. The hypothesis is that cording may have a vascular etiology

DETAILED DESCRIPTION:
Cords are bands of tissue that are present in the axilla following breast cancer surgery and may extend across the antecubital fossa and into the forearm. Cords are often painful to patients and limit their shoulder range of motion.The proposed study design involves the recruitment of patients who are enrolled in Partners Protocol # 2008P000540, a prospective analysis of symptoms, functionality and quality of life questionnaire to evaluate lymphedema in patients following treatment for breast cancer. This protocol recruits newly diagnosed breast cancer patients prior to any treatment interventions. Subjects are required to undergo volumetric arm measurements and complete the Lymphedema Evaluation Following Treatment for Breast Cancer Questionnaire (LEFT-BC) which will allow for the evaluation of changes in functionality, upper extremity utilization (fear associated avoidance), and quality of life. Throughout treatment patients will be screened before and after each treatment event: surgery, chemotherapy and radiation. Following the conclusion of treatment for breast cancer, patients will be measured at least 2 times per year (every 4-7 months). If during these study visits the patient notes cording symptoms, the research staff administering the questionnaire will be alerted. At this point, they will notify a designated medical provider who will perform a physical examination of the area to confirm the presence of cording. Once the presence of cording is verified, the patient will be provided with the opportunity to enroll in the proposed trial. Due to the current limited knowledge on the nature of the condition, the patients arm and axilla will have to be imaged within 7 days of the physical exam confirmation. The patients will be asked to return to the vascular imaging lab located on the Massachusetts's General Hospital's main campus. They will undergo a venous duplex ultrasound, on a General Electric LOGIQ-9 unit with a Phillips-IU-22 probe.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be enrolled in Partners protocol # 2008P000540 "Prospective Analysis of Symptoms, Functionality and Quality of Life Questionnaires to Evaluate Lymphedema in Patients Following Treatment for Breast Cancer"
* Confirmed case of cording by a medical provider (Physician, Nurse Practitioner, Physician Assistant)
* Participants must be at least 18 years of age
* Life expectancy of greater than 1 year.
* Ability to understand and the willingness to sign a written informed consent document.
* Willingness to comply with required follow up Perometer measurements and clinical visits.

Exclusion Criteria:

* Participants who are not enrolled or have been removed from Partners Protocol # 2008P000540 will be excluded from this trial.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of prior surgery or radiation to the head, neck, upper limb, or trunk.
* Patients with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The pathophysiology of cording following treatment for breast cancer | 7 days
  The cohort of 15 subject's images will be reviewed by the PI and a designated physician from the department of vascular medicine to determine if there is a vascular origin in the cords. Each image will be accessed for the following findings or involvement: Venous, lymphatic, fluid pockets, and striations on the cord.

SECONDARY OUTCOMES:
Cording and the onset of breast cancer related lymphedema | 30 days
  Subjects will be measured every 4-7 months with a perometer to determine if breast cancer related lymphedema is present.

CONTACTS AND LOCATIONS:
Overall Officials: Alphonse G Taghian, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States